CLINICAL TRIAL: NCT03399591
Title: Correlation Between Gait Disorders and Neuropsychological Profile in Patients With Alzheimer's Disease and Lewy Body Disease
Brief Title: Gait Disorders in Patients With Cognitive Decline
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6963
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-01

CONDITIONS: Gait Disorders, Neurologic
Keywords: Gait Disorders; Spatio-temporal parameters of walking; Alzheimer's disease; Lewy body disease
MeSH Terms: conditions — Gait Disorders, Neurologic; Mobility Limitation; Alzheimer Disease; Lewy Body Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevalence of neurodegenerative diseases will increase over the next decades driven by ageing population. It seems important to develop reliable, replicable and accessible diagnostic tools.

This is a prospective study whose objective is to study the spatio-temporal parameters of gait in patients with Alzheimer's and Lewy body diseases. 64 patients were included in this study. A comparison of the two pathologies was conducted, followed by an analysis based on four groups (mild, severe Alzheimer's disease, mild, severe Lewy body disease) and a study of the severity of the diseases. To study these parameters, we used the Gaitrite treadmill.

The analysis of spatio-temporal parameters of walking in Alzheimer's disease and Lewy body disease enables to identify discriminating variables between the two pathologies. The probability of suffering from an Alzheimer's disease decreases with the pace increase but increases with variations in length of the step, and with the rotation of the foot. While the probability of suffering from Lewy body disease increases with the pace, variations in the step duration, and the duration of double support.

These results are interesting but do not allow to establish a diagnostic score for these two diseases. The monitoring of the variations of these parameters at individual level would probably be more relevant and would enable to detect dual pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 50
* Hospitalized patient in day hospital
* Patient with an etiological diagnosis of his cognitive disorder
* Patient having a neuropsychological assessment
* Patient able to walk without technical help
* Patient having agreed to participate in the study

Exclusion Criteria:

- Refusal to participate in the study

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient over the age of 50 with a gait disorder
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
walking test | 1 hour after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Jérémie PERISSE, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Service de Gériatrie Hôpital de la Robertsau, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No